CLINICAL TRIAL: NCT01315483
Title: Diet Composition, Weight Control, and Breast Carcinogenesis
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Henry J. Thompson, Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CA125243
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; survivors; weight lose; dietary pattern
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low fat, high carb weight loss diet (Experimental): Ornish-like weight loss dietary pattern
  Interventions: Other: Weight Loss Dietary Pattern
- Low carb, high fat weight loss diet (Experimental): South-Beach-like weight loss diet pattern
  Interventions: Other: Weight Loss Dietary Pattern
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Weight Loss Dietary Pattern — Diet-physical activity program creating a weekly negative energy balance equivalent to 3500 kcal. Intervention groups receive PA protocol promoting the Physical Activity Guidelines and translated in step recommendations, but one of two diets with divergent dietary patterns (opposing fat and CHO content) that do not overlap >+5% in CHO and fat content. Macronutrient values reflect a 'pattern' or ratio within (LC 3:2 ratio for F:CHO; HC 1:4 ratio for F:CHO ) and between diets (LC:HC 3:1 for fat; LC:HC 1:2 for CHO). Six-week meal plans for five calorie levels available and incorporate educational material, supporting program components (e.g. self monitoring tools) and core competencies reinforcing weight loss behaviors in order to promote high levels of dietary adherence.
  Other Names: Low fat, high carb weight loss diet (Vivace Diet); Low carb, high fat weight loss diet (Ricca Diet)
  Arms: Low carb, high fat weight loss diet; Low fat, high carb weight loss diet

SUMMARY:
In the United States, overweight (BMI > 25 but < 30 Kg/m2) and obesity (BMI > 30Kg/m2) are increasing at epidemic rates. A significant association exists between being overweight or obese and breast cancer recurrence and survival. However, evidence continues to accumulate indicating that achieving or maintaining a healthy weight for height (Body Mass Index, BMI, 18.5-25Kg/m2) is associated with a reduced risk for breast cancer and with a decrease in breast cancer associated mortality. Despite this, there is a lack of randomized controlled trials exploring this association and how the process of fat loss or being successful in actually reaching a healthy weight for height differentially affects biomarkers for cancer recurrence.

Many dietary approaches for weight loss are currently available to the public, and each purports to offer advantages. However, there is little scientific evidence to indicate how these dietary approaches, some of which vary markedly in the foods that they limit or exclude, affect biomarkers for breast cancer risk. In particular, it is not know whether the critical factor in relation to weight and breast cancer is simply weight loss (negative energy balance), irrespective of the manner in which it is achieved, or if certain dietary approaches affect breast cancer risk biomarkers more favorably than others. Published data from our laboratory suggest that dietary pattern does matter, and therefore the goal of this study is to investigate the effects of two popular weight loss dietary approaches that differ in the extent to which they limit carbohydrate or fat consumption (with effects on dietary glycemic load) compared to a usual care group on prognostic markers for cancer recurrence in postmenopausal breast cancer survivors. The investigators hypothesize that in addition to the anticipated effects of fat loss on circulating levels of bioavailable sex steroid hormones, that the effects of excess fat on breast cancer prognosis can be attributed to three interrelated metabolic processes that affect cancer progression: altered glucose metabolism, chronic inflammation and excessive cellular oxidation.

DETAILED DESCRIPTION:
This study is designed to answer questions about how a dietary pattern either high or low in dietary carbohydrate and fat availability and fat loss influence metabolic and hormonal processes that may affect breast cancer recurrence. The investigators hypothesize that in addition to the anticipated effects of fat loss on circulating levels of bioavailable sex steroids, that the effects of excess fat on breast cancer prognosis can be attributed to three interrelated metabolic processes: altered glucose metabolism (IGF-1, IGFBP-3, glycated proteins), chronic inflammation (C-reactive protein, IL-6, TNF-alpha) and excessive cellular oxidation (8-hydroxy-2-deoxyguanosine and 8-isoprostane F-2 alpha).

A 6 month intervention study involving 370 post menopausal women who have been treated for breast cancer is proposed. Randomized women, stratified by resected stage, systemic adjuvant therapy and body mass index (> 25 and < 35 Kg/m2), will serve as either a non-intervention control group or will follow a tailored diet-physical activity program designed to create a weekly negative energy balance equivalent to 3500 kcal. The intervention groups will receive the same physical activity protocol, but one of two diets that differ in dietary pattern.

The specific aims are: Aim 1. Does a dietary pattern either high or low in available carbohydrate and fat alter the pattern of change observed in circulating factors involved in glucose homeostasis, chronic inflammation, cellular oxidation, and steroid hormone metabolism during progressive loss of body fat? The investigators will also examine how observed changes in these circulating factors related to changes indicators of breast cancer recurrence. Aim 2. Do circulating factors associated with glucose homeostasis, chronic inflammation, and cellular oxidation display the same pattern of change in response to progressive fat loss as circulating analytes associated with sex steroid metabolism? Analytes of interest will be measured monthly throughout the study. Aim 3. Does dietary glycemic load affect the magnitude or rate of fat loss? Plasma adipokines such as leptin and adiponectin and plasma ghrelin will be measured to provide biological determinants that may help explain differences in response.

The work proposed in this application should provide quantitative data about the importance of the magnitude of fat loss on metabolic and hormonal processes involved in cancer recurrence and provide guidance about effective dietary approaches that maximize weight loss benefits on breast cancer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivors
* Staged, resected breast cancer (> 4-months post radiation treatment, chemotherapy or surgery)
* Post-menopausal (no menses for > 6 months)
* No evidence of metastatic breast disease
* Willing to follow the diet plan prescribed
* Willing to follow the guidelines for alcohol consumption (no more than 1 standard alcoholic drink per day where one serving is defined as 12oz beer, 5 oz wine OR 1 oz hard liquor)
* Willing to maintain or increase current physical activity level
* Willing to wear a pedometer and keep a daily record of steps
* Willing to wear heart rate/ accelerometer device (Actiheart) continuously (24/7) for one week at the start and end of the study
* Willing to wear a body or swim suit and cap for body composition tests
* Willing to record food intake daily
* Willing to come to RMCC Rose for 11 individual and 5 group sessions over a 6 month period
* Willing to provide urine and fasting blood samples at 7 visits during the study
* Willing to make the commitment it takes to lose weight for the study
* Must have a Body Mass Index between 25Kg/m2 to 35Kg/m2.

Exclusion Criteria:

* Anticipates having surgery during the next 6 months
* Follows a special diet, e.g. gluten free, casein free, dairy free, vegetarian or other
* Lost 4 or more pounds during the previous month
* Taking weight loss medications during the study
* Being treated by a physician for diabetes
* Has an eating disorder
* Has digestive problems such as IBS (Irritable Bowel Syndrome), Crohn's or other
* Has had surgery involving constriction or removal of any portion of the gastrointestinal tract (gastric bypass, lap-band, bowel resection, colostomy etc.
* Diagnosed with hepatitis B, hepatitis C or HIV
* Has electronic devices implanted in their body (pacemaker, vagus nerve stimulator)
* Must not use any tobacco products

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-09; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Inflammation Markers | Baseline and montlhly for 6 months
  C-reactive protein, IL-6, TNF-alpha

SECONDARY OUTCOMES:
Body Fat Percentage (%) | Baseline and monthly for 6 months
  % Body fat, % lean muscle mass, Resting Metabolic Rate (RMR) using the BODPOD (Volumetric weighing; Life Measurement, Inc.) and Tanita Bioelectrical Impedence (BI)
Waist Hip Ratio | Baseline and monthly for 6 months
  Calculated by measuring and dividing waist and hip circumferences
Weight | Baseline and monthly for 6 months
  Using 1) BODPOD (Life Measurement, Inc.) and 2) Tanita Bioelectrical Impedence Scale
Bioavailable sex steroid hormones | Baseline and monthly for 6 months
  estradiol, estrone, sex hormone binding globulin (SHBG)
Glucose metabolism | Baseline and monthly for 6 months
  glucose, insulin, IGF-1, IGFBP-3, glycated proteins (HbA1c)
Cellular oxidation | Baseline and monthly for 6 months
  8-hydroxy-2-deoxyguanosine, DNA damage sensitivity and repair and 8-isoprostane-F-2-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Henry J Thompson, PhD, Principal Investigator — Colorado State University; Scot M Sedlacek, MD, Principal Investigator — Rocky Mountain Cancer Center
Locations (1):
- Rocky Mountain Cancer Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Thompson HJ, Sedlacek SM, Playdon MC, Wolfe P, McGinley JN, Paul D, Lakoski SG. Weight loss interventions for breast cancer survivors: impact of dietary pattern. PLoS One. 2015 May 26;10(5):e0127366. doi: 10.1371/journal.pone.0127366. eCollection 2015. PMID 26010254